CLINICAL TRIAL: NCT00389870
Title: A Randomised Clinical Trial of Treatment for Fluorouracil-Resistant Advanced Colorectal Cancer Comparing Standard Single-Agent Irinotecan Versus Irinotecan Plus Panitumumab and Versus Irinotecan Plus Ciclosporin [Panitumumab, Irinotecan & Ciclosporin in COLOrectal Cancer Therapy (PICCOLO)]
Brief Title: Irinotecan With or Without Panitumumab or Cyclosporine in Treating Patients With Advanced or Metastatic Colorectal Cancer That Did Not Respond to Fluorouracil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000510284; CTRU-PICCOLO-MO-05-7289; EUDRACT-2005-003492-20; CTAAC-CTRU-PICCOLO-MO-05-7289; AMGEN-CTRU-PICCOLO-MO-05-7289; EU-20647
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Cyclosporine; Irinotecan

INTERVENTIONS:
Biological: panitumumab
Drug: cyclosporine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cyclosporine may help irinotecan work better by making tumor cells more sensitive to the drug. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Panitumumab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether irinotecan is more effective when given with or without panitumumab or cyclosporine in treating colorectal cancer.

PURPOSE: This randomized phase III trial is studying irinotecan to compare how well it works when given with or without panitumumab or cyclosporine in treating patients with advanced or metastatic colorectal cancer that did not respond to fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy and toxicity of single-agent irinotecan hydrochloride (Ir) vs Ir with cyclosporine (IrC) in patients with fluorouracil-resistant advanced colorectal cancer.
* Compare the efficacy of single-agent Ir vs Ir with panitumumab (IrP) in these patients.

Secondary

* Correlate the toxicity of Ir and/or IrC with genetic variability in the enzymes involved in irinotecan hydrochloride's disposition pathway.
* Compare IrC to Ir and its metabolites (SN38; SN38G), in terms of pharmacokinetic profile.
* Correlate the benefit of IrP with tumor expression of epidermal growth factor receptor (EGFR) or its known down-stream molecules as a predictive measure.
* Correlate IrP efficacy or toxicity (specifically the severity of skin rash) with somatic alterations in the EGFR gene and/or with germline variability in related genes.

OUTLINE: This is a randomized, open-label, controlled, multicenter study. Patients are stratified according to prior cetuximab (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive irinotecan hydrochloride IV over 30-90 minutes on day 1.
* Arm II: Patients receive irinotecan hydrochloride IV over 15-40 minutes on day 1 and oral cyclosporine three times a day on days 1-3.
* Arm III: Patients receive panitumumab IV over 30-90 minutes followed by irinotecan hydrochloride IV over 30-90 minutes on day 1. Single-agent panitumumab may be continued during breaks in chemotherapy treatment.

In all arms, treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue treatment in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at 12 and 24 weeks.

After completion of study treatment, patients are followed every 12 weeks for 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,269 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma meeting 1 of the following criteria:

  * Previous or current histologically confirmed primary adenocarcinoma of the colon or rectum and clinical/radiological evidence of advanced or metastatic disease
  * Histologically or cytologically confirmed metastatic adenocarcinoma with clinical or radiological evidence of colorectal primary tumor
* Unidimensionally measurable disease
* Disease progression during or after prior fluorouracil with or without oxaliplatin therapy and/or with or without bevacizumab

  * Adjuvant therapy and/or prior therapy for advanced disease allowed
* No clinical or radiological evidence of pleural effusion or ascites causing ≥ grade 2 dyspnea
* No clinical or radiological evidence of biliary obstruction
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* Hemoglobin > 10.0 g/dL
* WBC > 3,000/mm³
* Platelet count > 100,000/mm³
* Glomerular filtration rate > 50 mL/min OR EDTA clearance > 60 mL/min
* Bilirubin < 1.46 mg/dL
* Alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* No history of Gilbert's syndrome
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Capable of completing quality of life questionnaires
* No prior anaphylactic allergic reaction to cetuximab
* No other prior or concurrent cancer (excluding nonmelanomatous skin cancer)
* No unresolved bowel obstruction, uncontrolled gastrointestinal infection, chronic enteropathy (e.g., Crohn's disease or ulcerative colitis), or chronic diarrhea (≥ 4 stools per day) of any cause
* No recent history of seizures
* No clinical or radiological evidence of interstitial pneumonitis or pulmonary fibrosis,
* Capable of reliable oral self-medication
* No other condition that would make the patient unsuitable for participation in this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No major thoracic or abdominal surgery within the past 4 weeks
* No systemic anticancer therapy within the past 3 weeks
* No prior irinotecan hydrochloride
* No grapefruit juice within 3 days before and after each chemotherapy treatment
* No experimental drug therapy or antibody therapy, other than cetuximab, within the past 6 weeks
* No systemic chemotherapy and/or cetuximab within the past 3 weeks
* No antifungals or antibiotics within the past 5 days
* No ongoing requirement for cyclosporine or any other medication including, but not limited to, the following:

  * Ketoconazole, fluconazole, itraconazole
  * Erythromycin, clarithromycin, norfloxacin
  * Diltiazem hydrochloride, verapamil, amiodarone hydrochloride
  * Fluvoxamine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
Proportion of patients treated with irinotecan hydrochloride (Ir) alone vs Ir and cyclosporine (IrC) who are progression-free at 12 weeks
Overall survival of patients treated with Ir vs Ir and panitumumab (IrP) and no prior cetuximab

SECONDARY OUTCOMES:
Proportion of patients free from treatment failure at 12 weeks in patients treated with Ir vs IrC
Overall survival in patients treated with Ir vs IrC
Nurse-assessed toxicity (all-cause mortality, diarrhea ≥ grade 3 at 12 weeks) in patients treated with Ir vs IrC
Progression-free at 12 weeks in patients treated with Ir vs IrP and no prior cetuximab
Nurse assessed toxicity (all-cause mortality) in patients treated with Ir vs IrP and no prior cetuximab
Progression-free survival in patients treated with Ir vs IrP and prior cetuximab
Best response at 1 year in patients treated with Ir vs IrP and prior cetuximab
Patient-assessed symptom/quality of life/acceptability scores at 12 and 24 weeks in patients treated with Ir vs IrP and prior cetuximab

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Seymour, MA, MD, FRCP, Study Chair — Cookridge Hospital
Locations (33):
- United Kingdom (33):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Eastbourne District General Hospital, Eastbourne, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - Airedale General Hospital, Keighley, England
  - Cookridge Hospital, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - UCL Cancer Institute, London, England
  - Queen Elizabeth Hospital - Woolwich, London, England
  - St. Mary's Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - South Tyneside District Hospital, South Shields, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales

REFERENCES:
- [Result] Seymour MT, Brown SR, Middleton G, Maughan T, Richman S, Gwyther S, Lowe C, Seligmann JF, Wadsley J, Maisey N, Chau I, Hill M, Dawson L, Falk S, O'Callaghan A, Benstead K, Chambers P, Oliver A, Marshall H, Napp V, Quirke P. Panitumumab and irinotecan versus irinotecan alone for patients with KRAS wild-type, fluorouracil-resistant advanced colorectal cancer (PICCOLO): a prospectively stratified randomised trial. Lancet Oncol. 2013 Jul;14(8):749-59. doi: 10.1016/S1470-2045(13)70163-3. Epub 2013 May 29. PMID 23725851
- [Result] Middleton G, Brown S, Lowe C, Maughan T, Gwyther S, Oliver A, Richman S, Blake D, Napp V, Marshall H, Wadsley J, Maisey N, Chau I, Hill M, Gollins S, Myint S, Slater S, Wagstaff J, Bridgewater J, Seymour M. A randomised phase III trial of the pharmacokinetic biomodulation of irinotecan using oral ciclosporin in advanced colorectal cancer: results of the Panitumumab, Irinotecan & Ciclosporin in COLOrectal cancer therapy trial (PICCOLO). Eur J Cancer. 2013 Nov;49(16):3507-16. doi: 10.1016/j.ejca.2013.06.017. Epub 2013 Aug 13. PMID 23953030
- [Result] Seligmann JF, Elliott F, Richman SD, Jacobs B, Hemmings G, Brown S, Barrett JH, Tejpar S, Quirke P, Seymour MT. Combined Epiregulin and Amphiregulin Expression Levels as a Predictive Biomarker for Panitumumab Therapy Benefit or Lack of Benefit in Patients With RAS Wild-Type Advanced Colorectal Cancer. JAMA Oncol. 2016 May 1;2(5):633-642. doi: 10.1001/jamaoncol.2015.6065. PMID 26867820